CLINICAL TRIAL: NCT05726071
Title: Electrocardiograph Changes and Holter Abnormalities in Children With Predialytic Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Wethab Khaled Mohamed, Pediatric resident at El Helal Hospital, Sohag University
Other Study IDs: Soh-med-23-01-12
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Predialytic Chronic Kidney Disease
Keywords: Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Holter — 24 hour electrocardiography
  Other Names: ECG Fukuda Denshi CardiMax ECG device model FCP-7101

SUMMARY:
CKD is a strong risk factor for cardiovascular disease and mortality , As in adults, cardiovascular disease occurs in some children with CKD before they reach ESRD as well as after

DETAILED DESCRIPTION:
This work aims to study the electrophysiological changes in cardiovascular system in children with predialytic CKD. ECG is important in detection of cardiac rhythm abnormalities, cardiac conduction defects and detection of myocardial ischemia

ELIGIBILITY:
Inclusion Criteria:

Age 1 to 15 year children with predialytic chronic kidney disease GFR.>15 ml\min per 1.73m2 , stages 1, 2, 3, 4 according to (KDOQI stages).

Exclusion Criteria:

* Age >15 year On regular dialysis GFR<15 ml\min per 1.73m2, Stage 5 according to (KDOQI stages). Children with known cardiovascular disease or known arrhythmia Patients on the potential medication affecting ECG result as B-blocker, antipsychotics , antidepressant

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with predialytic chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | One year
  Sinus tachycardia or bradycardia
changes in QT interval | One year
  Prolonged QT interval in ECG
QRS duration | One year
  Increase or decrease in ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

REFERENCES:
- [Background] Shafi S, Saleem M, Anjum R, Abdullah W, Shafi T. ECG Abnormalities In Patients With Chronic Kidney Disease. J Ayub Med Coll Abbottabad. 2017 Jan-Mar;29(1):61-64. PMID 28712176
- [Background] Park S, Yum Y, Cha JJ, Joo HJ, Park JH, Hong SJ, Yu CW, Lim DS. Prevalence and Clinical Impact of Electrocardiographic Abnormalities in Patients with Chronic Kidney Disease. J Clin Med. 2022 Sep 15;11(18):5414. doi: 10.3390/jcm11185414. PMID 36143060
- [Background] Chavers BM, Herzog CA. The spectrum of cardiovascular disease in children with predialysis chronic kidney disease. Adv Chronic Kidney Dis. 2004 Jul;11(3):319-27. doi: 10.1053/j.arrt.2004.04.002. PMID 15241746